CLINICAL TRIAL: NCT05098782
Title: Maintaining Behavior Change: A 6-year Follow-up of Adolescent 'Night-owls'
Status: Completed | Type: Observational
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor of clinical psychology, University of California, Berkeley
Other Study IDs: 2020-06-13428
Record Dates: First submitted 2021-10-12; First posted 2021-10-28 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Circadian Dysregulation
Keywords: Risk: Emotional, Cognitive, Behavioral, Social, Physical
MeSH Terms: conditions — Chronobiology Disorders; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A follow-up of a cohort of participants recruited for a prior study will be conducted. In the prior study, 10-18 years olds were provided one of two treatments to improve the sleep of adolescent night-owls. The follow-up will be approximately 6-years following participation in the prior study. The goal is to establish long-term outcomes in sleep and circadian functioning, in the five health-relevant domains and in engagement in sleep health behavior.

DETAILED DESCRIPTION:
A follow-up of a cohort of participants recruited for a prior study will be conducted. In the prior study, 10-18 years olds were provided one of two treatments to improve the sleep of adolescent night-owls. This follow-up will be conducted approximately 6-years following participation in the prior study. The participants will be 18-28 years of age.

Specific Aim 1: At the 6-year follow-up, participants recruited for the prior study will be assessed for sleep and circadian functioning and functioning in five health- relevant domains.

Specific Aim 2: The sample will also be assessed for their engagement in sleep health behavior.

This research will advance knowledge on: (a) longer-term outcomes and (b) the role of eveningness as a mechanism contributing to poorer outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria is individuals who participated in a previously-funded behavioral intervention (R01HD071065).

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be individuals who participated in a prior treatment study. They will be aged 18 and over.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Composite Scale of Morningness | 6 years
  Sum of 13-item; Mix of 4-point and 5-point response scale. Scores can range from 13 (extreme evening) to 55 (extreme morning).
Patient-Reported Outcomes Measurement Information System - Sleep Related Impairment | 6 years
  Sum of 8-items rated on a 5-point response scale. Scores can range from 8 to 40 (Higher score means more Sleep Related impairment)
Patient-Reported Outcomes Measurement Information System - Sleep Disturbance | 6 years
  Sum of 8-items rated on a 5-point response scale. Scores can range from 8 to 40 (Higher score means more Sleep Disturbance)
Youth Self-Report Composite Score for Emotional domain | 6 years
  A score of Depression, Anxiety, and Stress Scale (DASS) - Sum of 21 item scale, ranging 0-3. Scores can range from 0 to 63 (Higher score means worse outcome).
Youth Self-Report Score for Cognitive Domain | 6 years
  (Not a scale). A composite score of the Patient-Reported Outcomes Measurement Information System -Cognitive Function and the Patient-Reported Outcomes Measurement Information System-Cognitive Function - Abilities will be used to assess functioning in the Cognitive domain
Youth Self-Report Score for Behavioral Domain | 6 years
  (Not a scale) A composite score of the Brief Sensation Seeking Scale, Patient-Reported Outcomes Measurement Information System -Alcohol Use, Patient-Reported Outcomes Measurement Information System-Severity of Substance Use will be used to assess functioning in the Behavioral domain
Youth Self-Report Score for Social Domain | 6 years
  (Not a scale) A composite score of the Patient-Reported Outcomes Measurement Information System-Companionship, Patient-Reported Outcomes Measurement Information System-Emotional Support, Patient-Reported Outcomes Measurement Information System-Social Isolation, and Patient-Reported Outcomes Measurement Information System-Ability to Participate will be used to assess functioning in the Social domain.
Youth Self-Report Score for Physical Domain | 6 years
  (Not a scale) A composite score of the Modifiable Activity Questionnaire and Physical Health Questionnaire will be used to assess functioning in the Social domain.
Utilization Scale | 6 years
  14-item; 0-4 scale. Scores can range from 0 to 56 (Higher score means more utilization).
Self-Report Behavioral Automaticity Index integrated with the Utilization Scale | 6 years
  14-item; 0-4 scale. Scores can range from 0 to 56 (Higher score means more automaticity in utilization).

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 6 years
  19-item. First four items are integer responses. The rest of the items are on a 0-3 scale. Creates 7 composite scores, with the sum of the composite scores ranging from 0 to 21. (Higher score means increased severity of difficulty in all sleep area components).
Sleep Diary | 6 years
  (Not a scale) Night-to-night variability in the mid-point of sleep
Actigraphy | 6 years
  (Not a scale) Night-to-night variability in the mid-point of sleep
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Emotional Domain | 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Cognitive Domain | 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Behavioral Domain | 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Social Domain | 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Physical Domain | 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Composite Sleep Health Score | 6 years
  Composite Sleep Health Score which is defined as the sum of scores on 6 sleep health dimensions: Regularity (Midpoint fluctuation), Satisfaction (Sleep quality question on PROMIS-SD), Alertness (Daytime sleepiness question on PROMIS-SRI), Timing (Mean midpoint), Efficiency (Sleep efficiency) and Duration (Total Sleep Time). The Sleep Health Composite was constructed such that higher score indicates better sleep health.

OTHER OUTCOMES:
Change in Composite Scale of Morningness (CSM) | Baseline and at 6 years
  Sum of 13-item; Mix of 4-point and 5-point response scale. Scores can range from 13 (extreme evening) to 55 (extreme morning).
Change in Patient-Reported Outcomes Measurement Information System - Sleep Related Impairment | Baseline and at 6 years
  Sum of 8-items rated on a 5-point response scale. Scores can range from 8 to 40 (Higher score means more Sleep Related impairment)
Change in Patient-Reported Outcomes Measurement Information System - Sleep Disturbance | Baseline and at 6 years
  Sum of 8-items rated on a 5-point response scale. Scores can range from 8 to 40 (Higher score means more Sleep Disturbance)
Change in Depression, Anxiety, and Stress Scale (DASS) | Baseline and at 6 years
  Sum of 21 item scale, ranging 0-3. Scores can range from 0 to 63 (Higher score means worse outcome).
Change in Patient-Reported Outcomes Measurement Information System -Cognitive Function | Baseline and at 6 years
  Sum of 6-item; 5-point response scale. Scores can range from 6 to 30 (Higher score means higher cognitive function ).
Change in Patient-Reported Outcomes Measurement Information System-Cognitive Function - Abilities | Baseline and at 6 years
  Sum of 6-item; 5-point response scale. Scores can range from 6 to 30 (Higher score means higher cognitive function and abilities).
Change in Brief Sensation Seeking Scale | Baseline and at 6 years
  8-item; 5-point response scale; Scores can range from 8 to 40 (Higher score means higher sensation seeking).
Change in Patient-Reported Outcomes Measurement Information System -Alcohol Use | Baseline and at 6 years
  Sum of 7-item; 5-point response scale. Scores can range from 7 to 35 (Higher score means higher alcohol use).
Change in Patient-Reported Outcomes Measurement Information System -Severity of Substance Use | Baseline and at 6 years
  Sum of 7-item; 5-point response scale. Scores can range from 7 to 35 (Higher score means higher severity of substance use).
Change in Patient-Reported Outcomes Measurement Information System - Companionship | Baseline and at 6 years
  Sum of 4-item; 5-point response scale. Scores can range from 4 to 20 (Higher score means higher reported companionship).
Change in Patient-Reported Outcomes Measurement Information System - Emotional Support | Baseline and at 6 years
  Sum of 4-item; 5-point response scale. Scores can range from 4 to 20 (Higher score means higher reported emotional support).
Change in Patient-Reported Outcomes Measurement Information System - Social Isolation | Baseline and at 6 years
  Sum of 4-item; 5-point response scale. Scores can range from 4 to 20 (Higher score means higher levels of social isolation).
Change in Patient-Reported Outcomes Measurement Information System - Ability to Participate in Social Roles & Activities | Baseline and at 6 years
  Sum of 4-item; 5-point response scale. Scores can range from 4 to 20 (Higher score means higher ability to participate in Social Roles & Activities).
Change in Modifiable Activity Questionnaire | Baseline and at 6 years
  20-item. Scored by hours per week values and by Metabolic values.
Change in Physical Health Questionnaire | Baseline and at 6 years
  Sum of 15-item, 0-2 response scale. Scores can range from 0 to 30 (Higher score means worse physical symptoms)
Height | Baseline and at 6 years
  Centimeters (cm)
Weight | Baseline and at 6 years
  Pounds (lbs)
Hip circumference | Baseline and at 6 years
  Centimeters (cm)
Waist Circumference | Baseline and at 6 years
  Centimeters (cm)
Change in Utilization Scale | Baseline and at 6 years
  14-item; 1-5 scale. Scores can range from 14 to 70 (Higher score means more automaticity in utilization)
Sleep Diary | Baseline and at 6 years
  (Not a scale) Consensus sleep diary variables calculated separately for weekdays and weekends
Actigraphy | Baseline and at 6 years
  (Not a scale) Sleep parameters will be calculated separately for weekdays and weekends
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Emotional Domain | Baseline and at 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Cognitive Domain | Baseline and at 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Behavioral Domain | Baseline and at 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Social Domain | Baseline and at 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Youth Ecological Momentary Assessment Composite Risk Score of Functioning - Physical Domain | Baseline and at 6 years
  (Not a scale) Measured via Ecological Momentary Assessment
Alexian Brothers Urge to Self Injure Scale | 6 years
  5-item. 0-6 point scale. Total scores can range from 0-30 (Higher Score means higher Suicidal ideation)
Composite Sleep Health Score | Baseline and at 6 years
  Composite Sleep Health Score which is defined as the sum of scores on 6 sleep health dimensions: Regularity (Midpoint fluctuation), Satisfaction (Sleep quality question on PROMIS-SD), Alertness (Daytime sleepiness question on PROMIS-SRI), Timing (Mean midpoint), Efficiency (Sleep efficiency) and Duration (Total Sleep Time). The Sleep Health Composite was constructed such that higher score indicates better sleep health.
Sussex-Oxford Compassion Scale (SOCS) | Baseline and at 6 years
  Sum of 20-item, 5-point response scale. Scores can range from 20 to 100 (Higher score means higher compassion for self).
  Sub-scale items included.
Suicidal Behavior Questionnaire - Revised | 6 years
  4-item. Total scores can range from 3-18 (Higher Score means higher Suicidal ideation)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Background] Harvey AG, Hein K, Dolsen EA, Dong L, Rabe-Hesketh S, Gumport NB, Kanady J, Wyatt JK, Hinshaw SP, Silk JS, Smith RL, Thompson MA, Zannone N, Blum DJ. Modifying the Impact of Eveningness Chronotype ("Night-Owls") in Youth: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2018 Oct;57(10):742-754. doi: 10.1016/j.jaac.2018.04.020. Epub 2018 Aug 15. PMID 30274649
- [Derived] Susman ES, Patino EO, Tiab SS, Dong L, Gumport NB, Sarfan LD, Hinshaw SP, Harvey AG. Transdiagnostic Sleep and Circadian Intervention in Youth: Long-Term Follow-Up of a Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2025 Mar;64(3):362-374. doi: 10.1016/j.jaac.2024.05.001. Epub 2024 May 8. PMID 38729603